CLINICAL TRIAL: NCT04837599
Title: Artificial Intelligence Performance in Colonoscopy in Daily Practice: Randomised, Comparative Study of Pentax i10 Colonoscopes With or Without Endocuff Combined With Discovery™ or Without
Brief Title: Artificial Intelligence Performance in Colonoscopy in Daily Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gastroenterologie Baden-Wettingen (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Geyer Martin, Dr med. Geyer Martin, Principal investigator, Gastroenterologie Baden-Wettingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Gastro BW 1
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Colonic Polyp; Adenoma
Keywords: artificial intelligence
MeSH Terms: conditions — Colonic Polyps; Adenoma | interventions — Colonoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pentax i 10 (No Intervention): Patient gets normal colonoscopy without Endocuff or activation of artifical intelligence
- Pentax i 10 with artificial intelligence Discovery TM (Active Comparator): Normal Pentax i 10 colonoscope with on the special monitor acitvated artificial intelligence
  Interventions: Device: Discovery TM of Pentax medical on/off in colonoscopy
- Pentax i 10 with Endocuff TM (Active Comparator): Endocuff cap is mounted on the tip of the endoscope a cheap assistance device proven in former studies to increase adenoma detection rate.
  Interventions: Device: Discovery TM of Pentax medical on/off in colonoscopy
- Pentax i 10 with Endocuff TM and artificial intelligence Discovery TM (Active Comparator): Endocuff cap is mounted on the tip of the endoscope and artificial intelligence is activated on the monitor. hypothesis is that probably artificial intelligence and Endocuff combined potentiate their effect.
  Interventions: Device: Discovery TM of Pentax medical on/off in colonoscopy

INTERVENTIONS:
Device: Discovery TM of Pentax medical on/off in colonoscopy — on the monitor artificial integlligence Discovery can be switched on or off.
  Other Names: Endocuff mounted yes/no
  Arms: Pentax i 10 with Endocuff TM; Pentax i 10 with Endocuff TM and artificial intelligence Discovery TM; Pentax i 10 with artificial intelligence Discovery TM

SUMMARY:
randomized, controlled single center, single investigator study mainly in colorectal screening population in daily practice with and without artificial intelliegence (AI) named DiscoveryTM from Pentax medical. Patient randomly are allocated to one of four groups: Pentax i10 colonoscopes without any additional device, Pentax i 10 with DiscoveryTM (AI), Pentax i 10 with EndocuffTM and Pentax i10 with EndocuffTM and DiscoveryTM (AI).

The different groups are compared in terms of the different parameters: e.g. time of endoscopy, polyps (PDR) and adenoma detected (ADR).

DETAILED DESCRIPTION:
From August 2021 through August 2022 all patients undergoing a colonoscopy in a gastroenterologist's private practice are assigned using randomization tables to one or the other above mentioned groups. Time of the endoscopy (ascent, descent and intervention time), polyps detected and their histology are written down real time with a tablet computer anonymized with the patient number. Furthermore dosage of sedatives and over all satisfaction is traced.

1. endpoint is time gain in the different phase of the colonoscopy
2. endpoint is adenoma detection rate (ADR)

ELIGIBILITY:
Inclusion Criteria:

* all patients referred and fit for an ambulant colonoscopy

Exclusion Criteria:

* none

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Endoscopy time | within 45 minutes of examination
  measurement of ascent, descent and intervention time during colonoscopy

SECONDARY OUTCOMES:
polyp and adenoma detetction rate PDR and ADR | within 45 minutes of examination
  counts of polypes and their location in the colon and their histology

OTHER OUTCOMES:
Medication dosage | withn 45 minutes of examination
  Dosage of Propofol and Buscopan

CONTACTS AND LOCATIONS:
Locations (1):
- Martin Geyer, Wettingen, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No